CLINICAL TRIAL: NCT01639482
Title: Neuroimaging Studies of the Treatment of Bipolar Depression With Citalopram
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Darin Dougherty, Director, Division of Neurotherapeutics, Massachusetts General Hospital
Other Study IDs: 2009P002712
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Citalopram: Patients with bipolar disorder
- Placebo: Patients with bipolar disorder

SUMMARY:
Regional metabolic changes associated with response to 6 weeks of citalopram treatment, using 18-Fluorodeoxyglucose Positron Emission Tomography imaging, will be characterized (FDG PET).

DETAILED DESCRIPTION:
Regional metabolic changes associated with response to 6 weeks of citalopram treatment, using 18-Fluorodeoxyglucose Positron Emission Tomography imaging, will be characterized (FDG PET). The following hypothesis will be tested: Antidepressant response or remission in depressed BPD patients will be associated with changes in cortical (prefrontal, parietal, premotor) and paralimbic (hippocampus, anterior cingulate, subgenual cingulate, posterior cingulate, and anterior insula) regions, consistent with SRI antidepressant response in unipolar depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* Current age 18-64 years; DSM-IV diagnosis of BPD, type-I, or type-II; Enrolled in the Citalopram Study at Tufts Medical Center

Exclusion Criteria:

* Current pregnancy, or inability to utilize contraception, The presence of any metallic implants, History of claustrophobia

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with Bipolar Depression
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
rCMRglu | pre and post-treatment
  regional glucose metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Darin D Dougherty, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital - East, Charlestown, Massachusetts, United States